CLINICAL TRIAL: NCT05652387
Title: Preparing for Parenthood: A Father Inclusive Model of Prenatal Care
Brief Title: Father Inclusive Prenatal Care Study
Acronym: FIPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other); University of Wisconsin, Milwaukee (Other); Skills for Chicagoland's Future-Chicago (Unknown); Parent Child Center (PCC) Community Wellness Center (Unknown); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20062803-IRB01
Record Dates: First submitted 2022-11-21; First posted 2022-12-15 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Antenatal Care; Pregnancy Related; Parent-Child Relations; Parenting; Education; Counseling
Keywords: fatherhood; prenatal care; coparenting; parenting education

STUDY DESIGN:
Intervention Model Description: Descriptive/Evaluative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Father Inclusive Prenatal Care (Other): Co parenting, parenting education, employment and educational readiness training and support.
  Interventions: Behavioral: Father Inclusive Prenatal Care

INTERVENTIONS:
Behavioral: Father Inclusive Prenatal Care — Pregnant and parenting couples participate in co-parenting and parenting education, and job skills and education readiness

SUMMARY:
Young families need additional institutional support to help them meet the challenges of parenthood. Prenatal clinics are well situated to address some of their needs by expanding services to include fathers. The Father Inclusive Prenatal Care (FIPC) model is designed to prepare young men for the challenges of parenting by supporting the development of their relationship skills as part of routine prenatal healthcare. This approach involves assessing expectant fathers and mothers with a "parent prep-check" (PPC) to identify their needs and then offer services to address those needs and prepare them for parenthood. Services include: (1) parent education about how to understand and care for infants, and how to build secure parent-child bonds; (2) an evidence-based co-parenting program to strengthen and stabilize their family; and (3) educational and employment support designed to help young parents find and keep living wage jobs. The project will be implemented through several community based healthcare sites that are well positioned to engage young fathers through their prenatal clinics. To extend the reach and accessibility of the model, trainings and most services will be available online. As a result of participating in this project it is expected that young couples will have better co-parenting relationships and be better prepared to take care of their infants.

DETAILED DESCRIPTION:
Recruitment: This project will recruit/engage young expectant fathers using a multi-stage process. First, primary care providers (PCP) will ask their patients (17-25-year-old pregnant women) about the degree to which the father of her child will be participating in parenting and supporting their baby. If the mother anticipates the fathers' involvement, the provider will tell her about the Parent Prep-Checks (PPC), give her a brochure about describing that process (including incentives), and ask about connecting her with members of the research team in order to receive additional information. The research team members will establish father eligibility based upon age (18-29 years) and schedule time to meet with both parents.

The intake process - the Parent Prep Check - is a strategy for engaging young fathers and mothers in research and intervention activities. In addition to collecting useful baseline data, the PPC is designed to build a strong alliance between project staff and participants. For example, FIPC intake staff are trained to administer a semi-structured interview designed to help participants articulate their feelings about becoming parents, which most find to be an interesting and rewarding experience. Then to facilitate recruitment into the intervention, a motivational interviewing approach is used that (a) gives feedback to participants based on their self-reported data and (b) engages them in thinking about what services will help them get ready for parenthood. When fathers are given the chance to say what concerns them, they are more likely to be receptive to participating in programs that can address those concerns. Intake staff will then introduce expectant parents to a FIPC provider, who discusses the goals and benefits of the FIPC program. Emphasizing how FIPC programs address a parent's self-identified goals has been an effective way to engage and retain participants.

The most critical element in this process is the quality of communication between FIPC staff and the expectant mother and father. If done well, both parents will feel appreciated, supported, and respected. Another key factor is flexibility. FIPC staff are trained to be as accommodating as possible about scheduling appointments. Related to this, almost all FIPC services and research activities are available online to increase participant reach and accessibly.

Finally, fathers and mothers are told they will be reimbursed for their time. Incentivizing patients is not sustainable over the long run; however, it is deemed necessary to get a representative sample for this project. In years 4 and 5, incentives for services will be reduced as part of the sustainability plan. In past projects, this strategy has been effective in recruiting between 60 and 75% of eligible expectant fathers.

Staff at partner clinics and Rush program coordinators who will be trained on the FIPC program and research/evaluation data protocol will be responsible for recruiting the sample. The clinic staff will be asking eligible mothers if they think their partner (father of the baby) would be interested in participating. The FIPC program coordinators will be responsible for contacting fathers and recruiting them to participate after mothers share their contact information.

Barrier reduction strategies will be used to support participant engagement. Due to the length of the Parent Prep check (3 hours), expectant parents will be offered a snack during the interview.

ELIGIBILITY:
Inclusion Criteria:

* Women: pregnant woman
* Men & women have to be willing to participate at baseline interview together

Exclusion Criteria:

* Men & Women: Language other than Spanish or English and cognitive disability interfering with ability to understand the informed consent process.

Ages: 17 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women age 17-25 Expectant biological fathers age 18-29
Enrollment: 216 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Change in conflict in Adolescent Dating Relationship Inventory- Short Form | Change from Baseline (2nd trimester of pregnancy) at 6 months and 18 months post birth
  Used to measure couple relationships and potential conflict.
Parenting Stress Index - Short Form | At 6 months and 18 months post birth
  Evaluates parents' perception of parenting-related stress
Perceived Maternal Parenting Self-Efficacy Tool | Time 2 - six months post birth
  Evaluates how confident parents feel taking care of their infant
Self-efficacy for Parenting Task Index - Toddler-Short | Time 3 - eighteen months post birth
  Evaluates how capable parents feel of addressing their child's needs.
Julion Index of Paternal Involvement | At 6 months and 18 months post birth
  Measures how often fathers are involved with their children in a variety of activities
Brief Infant Toddler Social & Emotional Assessment (BITSEA) | Time 3- eighteen months post birth
  This form is used to measure infant social-emotional development
Quality of Relationship Inventory | At 6 months and 18 months post birth
  Examines the quality of the relationship between co-parenting couples

SECONDARY OUTCOMES:
Maternal Health Outcome Assessment | Six months post birth
  Instrument used to report infant birth and mother delivery data.
Trait Emotional Intelligence Questionnaire | At 6 months and 18 months post birth
  Measure of emotional intelligence
Parent Health Questionnaire (PHQ9) | At 6 months and 18 months post birth
  Screening for symptoms of depression

OTHER OUTCOMES:
Changes in Administration for Children & Families Survey | Change from baseline (2nd trimester of pregnancy) at 6 months and 18 months post birth.
  Detailed demographic information required by funder
Post-traumatic Stress Symptoms Questionnaire | At 6 months and 18 months post birth
  screens for post traumatic stress
The CRAFFT Screener for Drug and Alcohol Abuse Questionnaire | At 6 months and 18 months post birth
  Screens for substance abuse
Parent Readiness Questionnaire | Baseline (2nd trimester of pregnancy)
  Examines fathers readiness to be a parent

CONTACTS AND LOCATIONS:
Overall Officials: Wrenetha A Julion, PhD, MPH, RN, Principal Investigator — Rush University Medical Center; Paul w Florsheim, PhD, Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Based upon guidance by the funding agency de-identified descriptive and quantitative data will be housed at a designated site and made available to eligible researchers.
Supporting Information: Study Protocol, SAP
Time Frame: At the completion of the study following all analyses by the primary research team.
Access Criteria: All data will be deidentified; information will be provided about the type of data available; the research proposal of the requestor will be reviewed by an independent review panel; data will be available for use but not downloadable; registration and the use of data use agreements are required;

REFERENCES:
- [Background] Florsheim P, Burrow-Sanchez JJ, Minami T, McArthur L, Heavin S, Hudak C. Young parenthood program: supporting positive paternal engagement through coparenting counseling. Am J Public Health. 2012 Oct;102(10):1886-92. doi: 10.2105/AJPH.2012.300902. Epub 2012 Aug 16. PMID 22897540
- [Background] Florsheim, P., McArthur, L., Hudak, C., Heavin, S., & Burrow-Sanchez, J. (2011). The Young Parenthood Program: Preventing intimate partner violence between adolescent mothers and young fathers. Journal of Couple & Relationship Therapy, 10(2), 117-134.
- [Background] Paul, H. A. (2015). The Young Parenthood Program: A Guide to Helping Young Mothers and Fathers Become Effective Co-Parents, by P. Florsheim: New York, NY: Oxford University Press, vii+ 222 pp., $45.00 (paperback).
- [Background] Julion WA, Breitenstein SM, Waddell D. Fatherhood intervention development in collaboration with African American non-resident fathers. Res Nurs Health. 2012 Oct;35(5):490-506. doi: 10.1002/nur.21492. Epub 2012 Jun 8. PMID 22685066
- [Background] Julion WA, Sumo J, Bounds DT, Breitenstein SM, Schoeny M, Gross D, Fogg L. Study protocol for a randomized clinical trial of a fatherhood intervention for African American non-resident fathers: Can we improve father and child outcomes? Contemp Clin Trials. 2016 Jul;49:29-39. doi: 10.1016/j.cct.2016.05.005. Epub 2016 May 28. PMID 27241687
- [Background] Julion, W. A., Sumo, J. N., Schoeny, M. E., Breitenstein, S. M., & Bounds, D. T. (2021). Predictors of Maternal Participation in Fatherhood Intervention Research With African American Nonresident Fathers. Research on Social Work Practice, 10497315211005538.